CLINICAL TRIAL: NCT01222767
Title: Phase II Multicenter, Open-label, Clinical and Pharmacokinetic Study of Zalypsis® (PM00104) in Patients With Unresectable Locally Advanced and/or Metastatic Ewing Family of Tumors (EFT) Progressing After at Least One Prior Line of Chemotherapy
Brief Title: Study of Zalypsis® (PM00104) in Patients With Unresectable Locally Advanced and/or Metastatic Ewing Family of Tumors (EFT) Progressing After at Least One Prior Line of Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM104-B-003-10
Record Dates: First submitted 2010-10-08; First posted 2010-10-18 (Estimated); Results first posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-07

CONDITIONS: Ewing's Sarcoma; Primitive Neuroectodermal Tumor (PNET); Askin's Tumor of the Chest Wall; Extraosseous Ewing's Sarcoma (EOE)
Keywords: EFT; PNET; EOE
MeSH Terms: conditions — Sarcoma, Ewing; Neuroectodermal Tumors, Primitive | interventions — PM 00104

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Zalypsis

INTERVENTIONS:
Drug: Zalypsis — Zalypsis is provided as a lyophilized powder for concentrate for solution for infusion in a strength of 2.5 mg/vial.
  Other Names: PM00104

SUMMARY:
This is a phase II Multicenter, Open-label, Clinical and Pharmacokinetic Study of Zalypsis® (PM00104) in Patients with Unresectable Locally Advanced and/or Metastatic Ewing Family of Tumors (EFT) Progressing After at Least One Prior Line of Chemotherapy to determine the antitumor activity of Zalypsis.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent, obtained from the patient or his/her representative before the beginning of any specific study procedures.
2. Age ≥ 16 years.
3. Histologically or cytologically confirmed EFT (Ewing Family of Tumors), with recurrent disease.
4. Documented failure to at least one prior chemotherapy regimen for their disease.
5. Radiographic documentation of disease progression at study entry.
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score ≤ 2.
7. Life expectancy ≥ 3 months.
8. Complete recovery from the effects of drug-related adverse events (AEs) derived from previous treatments, excluding alopecia and grade 1 peripheral neuropathy, according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v. 4.0.
9. At least one measurable lesion ("target lesion" according to the RECIST v.1.1), located in a non-irradiated area and adequately measured less than four weeks before study entry. Tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is clearly documented or biopsy proven.
10. Absolute neutrophil count (ANC) ≥ 1.5 x 109/l; platelet count ≥ 100 x 109/l, and hemoglobin ≥ 9 g/dl.
11. Adequate renal function: calculated creatinine clearance (using Cockcroft and Gault's formula) ≥ 30 ml/min.
12. Adequate hepatic function:

    * Total bilirubin ≤ 1.5 x upper limit or normality (ULN), unless due to Gilbert's syndrome.
    * Alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤ 3 x ULN (≤ 5 x ULN in case of hepatic metastases), and alkaline phosphatase (AP) ≤ 2.5 x ULN (≤ 5 x ULN in case of extensive bone involvement).
    * Albumin ≥ 25 g/l.
13. Left ventricular ejection fraction (LVEF) within normal limits (LVEF of at least 50%).
14. Women of childbearing potential must have a negative serum pregnancy test before study entry. Both women and men must agree to use a medically acceptable method of contraception throughout the treatment period and for three months after discontinuation of treatment. Acceptable methods of contraception include complete abstinence, intrauterine device (IUD), oral contraceptive, subdermal implant and double barrier (condom with a contraceptive sponge or contraceptive suppository).

Exclusion Criteria:

1. Prior therapy with Zalypsis®.
2. Pregnant or lactating women or women of childbearing potential not using an appropriate contraceptive method.
3. Less than three weeks from prior radiation therapy, biological therapy or chemotherapy.
4. Less than six weeks from prior nitrosourea, mitomycin C, high-dose chemotherapy or radiotherapy involving the whole pelvis or over 50% of the spine, provided that acute effects of radiation treatment have resolved. Hormonal therapy and palliative radiation therapy (i.e., for control of pain from bone metastases) must be discontinued before study entry.
5. Patients with a prior invasive malignancy (except non-melanoma skin cancer and in situ cervix carcinoma) who have had any evidence of disease within the last five years or whose prior malignancy treatment contraindicates the current protocol therapy.
6. Evidence of progressive or symptomatic central nervous system (CNS) metastases or leptomeningeal metastases.
7. Other diseases or serious conditions:

   * Increased cardiac risk, as defined by:

     * Unstable angina or myocardial infarction within 12 months before inclusion in the study.
     * New York Heart Association (NYHA) grade II or greater congestive heart failure.
     * Symptomatic arrhythmia or any arrhythmia requiring ongoing treatment.
     * Abnormal electrocardiogram (ECG), i.e., patients with the following are excluded: QT prolongation - QTc > 480 msec; signs of cardiac enlargement or hypertrophy; bundle branch block; partial blocks; signs of ischemia or necrosis, and Wolff Parkinson White patterns.
     * History or presence of valvular heart disease.
     * Uncontrolled arterial hypertension despite optimal medical therapy.
     * Previous mediastinal radiotherapy.
     * Previous treatment with doxorubicin at cumulative doses exceeding 400 mg/m2.
   * History of significant neurological or psychiatric disorders.
   * Active infection requiring systemic treatment.
   * Significant non-neoplastic liver disease (e.g., cirrhosis).
   * Known hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
   * Immunocompromised patients, including those known to be infected with the human immunodeficiency virus (HIV).
   * Uncontrolled (i.e., requiring relevant changes in medication within the last month or hospital admission within the last three months) endocrine diseases (e.g., diabetes mellitus, hypo- or hyperthyroidism, adrenal disorder).
8. Any other major illness that, in the Investigator's judgment, will substantially increase the risk associated with the patient's participation in the study. The Investigator should feel free to consult the Study Coordinator or the Sponsor(s) in case of uncertainty in this regard.
9. Limitation of the patient's ability to comply with the treatment or to follow-up at a participating center. Patients enrolled into this trial must be treated and followed at a participating center.
10. Treatment with any investigational product within 30 days prior to inclusion in the study.
11. Known hypersensitivity to any component of Zalypsis®.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fariba Navid, MD, Principal Investigator — St. Jude Children 's Research Hospital; Sant P Chawla, MD, Principal Investigator — Sarcoma Oncology Center; Jean Yves Blay, MD, Principal Investigator — Centre Leon Berard; Stefano Ferrari, MD, Principal Investigator — Istituto Ortopedici Rizzoli; Armando Santoro, Prof., Principal Investigator — Istituto Clinico Humanitas; Paolo Casali, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano; Robin L. Jones, MD, Principal Investigator — Seattle Cancer Care Alliance
Locations (7):
- United States (3):
  - Sarcoma Oncology Center, Santa Monica, California
  - St. Jude Children 's Research Hospital, Memphis, Tennessee
  - Seattle Cancer Care Alliance, Seattle, Washington
- Centre Léon Bérard, Lyon, France
- Italy (3):
  - Istituto Ortopedici Rizzoli, Bologna
  - Istituto Nazionale dei Tumori, Milan
  - Istituto Clinico Humanitas, Rozzano

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 17 patients were included and 16 of them were treated with PM00104 at five investigational sites from the USA (n=3), France and Italy. The patients participated in this study between 22 December 2010 (first consent) and 21 May 2012 (last follow-up). First and last doses were administered on 4 January 2011 and 24 January 2012, respectively
Groups:
- PM00104: PM00104 was administered at a dose of 2 mg/m2 as a 1-hour i.v. infusion d1, d8 and d15 q4wk to patients with advanced and/or metastatic Ewing's sarcoma previously treated with at least one line of chemotherapy. A treatment cycle consisted of PM00104 administration on Days 1, 8 and 15, plus one week of follow-up. Study evaluations had to be completed during each cycle prior to subsequent PM00104 infusion. Treatment cycles were repeated every four weeks
Period: Overall Study
Arm/Group | PM00104
Started | 17
Received Treatment | 16
Completed | 0
Not Completed | 17
Not completed — Progressive disease | 13
Not completed — Adverse Event | 2
Not completed — Surgical resection | 1
Not completed — Never treated | 1

BASELINE CHARACTERISTICS:
Arm/Group | PM00104
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 13
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 23 [15 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12
  Italy | 3
  France | 2
ECOG PS [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group Performance Status, ECOG PS 0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours
  3. Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours
  4. Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair
  5. Dead
  Participants
    0 | 9
    1 | 7
    2 | 1
Tumor diagnosis [Count of Participants; unit: Participants]
  Ewing's bone sarcoma | 13
  Extraosseous sarcoma | 4
Primary location at diagnosis [Count of Participants; unit: Participants]
  Lower extremity | 7
  Trunk/abdominal wall | 7
  Upper extremity | 1
  Unknown | 2
Metastatic disease [Count of Participants; unit: Participants] | 17
Time from diagnosis to first infusion [Median (Full Range); unit: months] | 43.3 [13.8 to 81.3]
Time from last disease progression to first infusion [Median (Full Range); unit: months] | 0.3 [0.1 to 1.8]
Sites of disease at diagnosis [Count of Participants; unit: Participants]
  1 | 7
  2 | 6
  3 | 3
  >3 | 1
Prior radiotherapy [Count of Participants; unit: Participants] | 14
Prior Antitumor surgery (palliative or curative) [Count of Participants; unit: Participants] | 14
Prior Systemic anticancer therapy [Count of Participants; unit: Participants] | 17

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Overall response rate (ORR), defined as the percentage of patients with confirmed objective response (OR), either CR or PR according to the RECIST v.1.1.
  CR, complete response: disappearance of all lesions; PD, disease progression: ≥10% increase in target lesion size and does not meet tumor density criteria of PR density; PR, partial response: ≥10% decrease in target lesion size or ≥15% decrease in tumor density; SD, stable disease: none of the CR, PR, or PD criteria met; RECIST, Response Evaluation Criteria in Solid Tumors
Time Frame: At baseline and every other cycle (± 1 week) until evidence of PD, up to 2 years
Population: One patient never treated
Measure: Count of Participants; unit: Participants
Arm/Group | PM00104
Number analyzed (Participants) | 16
Participants | 0

2. Secondary Outcome: Best Tumor Response
Description: Best tumor response was defined as the best response achieved during the study according to RECIST v1.1 CR, complete response: disappearance of all lesions; PD, disease progression: ≥10% increase in target lesion size and does not meet tumor density criteria of PR density; PR, partial response: ≥10% decrease in target lesion size or ≥15% decrease in tumor density; SD, stable disease: none of the CR, PR, or PD criteria met; RECIST, Response Evaluation Criteria in Solid Tumors
Time Frame: At baseline and every other cycle (± 1 week) until evidence of PD, up to 2 years
Population: One patient never treated Two patients were non-evaluable for efficacy because they were withdrawn due to toxicity without any tumor assessment after the start of study treatment and were considered as "treatment failures"
Measure: Count of Participants; unit: Participants
Arm/Group | PM00104
Number analyzed (Participants) | 14
Participants
  SD | 4
  PD | 10

3. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS), defined as the time from the first day of study treatment to the day of negative assessment (progression or death), start of subsequent antitumor therapy, or last tumor evaluation.
  PD, disease progression: ≥10% increase in target lesion size and does not meet tumor density criteria of PR density; PR, partial response: ≥10% decrease in target lesion size or ≥15% decrease in tumor density
Time Frame: From the first day of study treatment to the day of negative assessment (progression or death), start of subsequent antitumor therapy, or last tumor evaluation, up to 2 years
Population: One patient never treated
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PM00104
Number analyzed (Participants) | 16
months | 1.8 [0.9 to 3.5]

4. Secondary Outcome: Progression-free Survival at 3 Months
Description: as for outcome 3
Time Frame: At 3 months
Population: One patient never treated
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PM00104
Number analyzed (Participants) | 16
percentage of participants | 28.6 [4.9 to 52.2]

5. Secondary Outcome: Overall Survival
Description: Overall survival (OS), defined as the time from the first day of treatment to the date of death (or the last day when the patient was known to be alive). Survival was to be followed for up to six months after the last treatment visit of the last patient, or 12 months after the last patient was included, whichever occurred first.
Time Frame: from the first day of treatment to the date of death, up to 2 years
Population: One patient never treated
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PM00104
Number analyzed (Participants) | 16
months | NA [NA to NA] — Median survival could not be calculated because more than half of patients were still living

6. Secondary Outcome: Overall Survival Rate at 6 Months
Description: as for outcome 5
Time Frame: At 6 months
Population: One patient never treated
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PM00104
Number analyzed (Participants) | 16
percentage of participants | 62.5 [38.8 to 86.2]

7. Secondary Outcome: Overall Survival Rate at 12 Months
Description: as for outcome 5
Time Frame: At 12 months
Population: One patient never treated
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PM00104
Number analyzed (Participants) | 16
percentage of participants | 54.7 [29.5 to 79.9]

8. Secondary Outcome: PM00104 Plasma PK Parameters (Cmax) at First Infusion
Description: Cmax Maximum plasma concentration, directly determined from the experimental data
Time Frame: 0 (Pre-infusion) and 5 min, 30 min, 2 hours, 6 hours, 24 hours, 48 hours and 168 hours after the end of first infusion (Day 1)
Population: Fourteen of the 16 patients treated in this study had plasma profiles
Measure: Mean (Standard Deviation); unit: μg/l
Arm/Group | PM00104
Number analyzed (Participants) | 14
μg/l | 21.23 (8.35)

9. Secondary Outcome: PM00104 Plasma PK Parameters (AUC) at First Infusion
Description: AUC Area under the plasma concentration-time curve from time zero to infinity
Time Frame: as for outcome 8
Population: Fourteen of the 16 patients treated in this study had plasma profiles
Measure: Mean (Standard Deviation); unit: h*μg/l
Arm/Group | PM00104
Number analyzed (Participants) | 14
h*μg/l | 87.06 (75.49)

10. Secondary Outcome: PM00104 Plasma PK Parameters (Cmax) at Second Infusion
Description: Cmax Maximum plasma concentration, directly determined from the experimental data
Time Frame: 0 (Pre-infusion) and 5 min, 30 min, 2 hours, 6 hours, 24 hours, 48 hours and 168 hours after the end of second infusion (Day 8)
Population: Eleven of the 16 patients treated in this study had plasma profiles at second infusion
Measure: Mean (Standard Deviation); unit: μg/l
Arm/Group | PM00104
Number analyzed (Participants) | 11
μg/l | 22.37 (8.77)

11. Secondary Outcome: PM00104 Plasma PK Parameters (AUC) at Second Infusion
Description: AUC Area under the plasma concentration-time curve from time zero to infinity
Time Frame: as for outcome 10
Population: Eleven of the 16 patients treated in this study had plasma profiles at second infusion
Measure: Mean (Standard Deviation); unit: h*μg/l
Arm/Group | PM00104
Number analyzed (Participants) | 11
h*μg/l | 69.76 (17.69)

ADVERSE EVENTS:
Time Frame: From first infusion to study termination, up to 2 years
Description: Sixteen of 17 patients included in this study were treated with PM00104 and were therefore evaluable for safety
Arm/Group | PM00104
All-Cause Mortality (participants affected / at risk) | 7/16
Serious Adverse Events (participants affected / at risk) | 2/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PM00104 (N=16)
Acute sinusitis (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PM00104 (N=16)
Anaemia (Blood and lymphatic system disorders) | 2 (4)
Neutropenia (Blood and lymphatic system disorders) | 7 (11)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Palpitations (Cardiac disorders) | 3 (3)
Pericardial effusion (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2)
Ear congestion (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Eye swelling (Eye disorders) | 1 (1)
Myopia (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (7)
Stomach discomfort (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Chest pain (General disorders) | 3 (3)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 7 (10)
Non-cardiac chest pain (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 6 (6)
Nasopharyngitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Breath sounds abnormal (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 2 (3)
Headache (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (10)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Oropharyngeal blistering (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Pallor (Vascular disorders) | 1 (1)
Superior vena caval occlusion (Vascular disorders) | 1 (2)
Venous thrombosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review.

DOCUMENTS (2):
  • Study Protocol (2010-07-30): https://cdn.clinicaltrials.gov/large-docs/67/NCT01222767/Prot_000.pdf
  • Statistical Analysis Plan (2013-02-07): https://cdn.clinicaltrials.gov/large-docs/67/NCT01222767/SAP_001.pdf